CLINICAL TRIAL: NCT05145621
Title: An Open-Label, Balanced, Randomized, 2-Treatment, 2-Sequence, 2-Period, Single Dose, Crossover Oral Bioequivalence Study of Two Formulations of Fingolimod Capsules (3 x 0.5 mg) in Healthy Adult Human Subjects Under Fasting Conditions
Brief Title: Oral Bio-equivalence Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alembic Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: AMC-P6-855
Record Dates: First submitted 2015-11-23; First posted 2021-12-06 (Actual); Last update posted 2021-12-21 (Actual); Status verified 2021-12

CONDITIONS: Bioequivalence; Safety
MeSH Terms: interventions — Fingolimod Hydrochloride

STUDY DESIGN:
Intervention Model Description: two way crossover
Oversight: Data Monitoring Committee: No

ARMS (2):
- Test (Active Comparator): Fingolimod 0.5 mg capsules - (administered as 3 x Fingolimod 0.5 mg capsules)
  Interventions: Drug: Fingolimod 0.5 mg capsules- Test drug
- Reference (Active Comparator): Fingolimod 0.5 mg capsules -(administered as 3 x Fingolimod 0.5 mg capsules)
  Interventions: Drug: Fingolimod 0.5 mg capsules- Test drug

INTERVENTIONS:
Drug: Fingolimod 0.5 mg capsules- Test drug — An oral dose of the assigned formulation (3 capsules) will be administered in the morning to subjects with about 240 mL of water at ambient temperature according to the randomization scheme.
  Other Names: Fingolimod 0.5 mg capsules- Reference drug

SUMMARY:
Title of Study: An Open-Label, Balanced, Randomized, 2-Treatment, 2-Sequence, 2-Period, Single Dose, Crossover Oral Bioequivalence Study of Two Formulations of Fingolimod Capsules (3 x 0.5 mg) in Healthy Adult Human Subjects Under Fasting Conditions.

Objective: The objective of this study is to compare the oral bioavailability and characterize the pharmacokinetic profile of the test formulation relative to that of reference formulation in healthy, adult, human subjects under fasting conditions and to assess the bioequivalence.

ELIGIBILITY:
Inclusion Criteria:

Volunteers meeting all of the following criteria will be considered for enrollment in the study:

1. Availability for the entire study period 2. Motivated volunteer and absence of intellectual problems likely to limit the validity of consent to participate in the study or the compliance with protocol requirements; ability to cooperate adequately; ability to understand and observe the instructions of the physician or designee 3. Male or female volunteer 4. A female volunteer must meet one of the following criteria:

1. Physiological postmenopausal status, defined as the following:

   1. no menses for at least one year (absence of menses should not be due to lactational amenorrhea); and
   2. FSH levels ≥ 40 mIU/mL at screening; or
2. Surgical postmenopausal status, defined as the following:

   1. bilateral oophorectomy; and
   2. absence of menses for at least 3 months; and
   3. FSH levels ≥ 40 mIU/mL at screening; or
3. Hysterectomy with FSH levels ≥ 40 mIU/mL at screening If the postmenopausal volunteer has an FSH of < 40 mIU/mL, but meets the above criteria in either (1), (2) or (3) and all the other inclusion criteria in section 5.2, the volunteer may be included in the study if the estradiol serum level measured at screening is equal to or below 150 pmol/L. In the case of hysterectomy, if FSH and estradiol do not meet the criteria, inclusion of the volunteer will be based on medical judgment. 5. Volunteer aged of at least 18 years but not older than 45 years 6. Volunteer with a BMI greater than or equal to 18.50 kg/m2 and below 30.00 kg/m2 7. Volunteer with a minimum body weight of at least 60 kg 8. Non- or ex-smokers; an ex-smoker being defined as someone who completely stopped smoking and/or using tobacco/tobacco-containing products for at least 6 months before day 1 of this study 9. Clinical laboratory values within the laboratory's stated normal range; if not within this range, they must be without any clinical significance 10. Have no clinically significant diseases captured in the medical history or evidence of clinically significant findings on physical examination and/or clinical laboratory evaluations (hematology, general biochemistry, ECG and urinalysis) 11. Willingness to adhere to the protocol requirements as evidenced by the informed consent form (ICF) duly read, signed and dated by the volunteer 12. Volunteer agrees not to participate in another clinical study for up to 10 weeks following the last drug administration The ICF must be signed by all volunteers prior to their participation in the study.

Exclusion Criteria:

Volunteers presenting any of the following will not be included in the study:

1. Difficulty donating blood
2. Difficulty swallowing solids like tablets or capsules
3. Seated pulse rate less than 60 bpm or more than 100 bpm at screening
4. History of significant hypersensitivity to fingolimod or any related products (including excipients of the formulations) as well as severe hypersensitivity reactions (like angioedema) to any drugs
5. Presence of significant gastrointestinal, liver or kidney disease, or any other conditions known to interfere with the absorption, distribution, metabolism or excretion of drugs or known to potentiate or predispose to undesired effects
6. History of significant gastrointestinal, liver or kidney disease that may affect drug bioavailability
7. History or presence of significant cardiovascular, respiratory, pulmonary, hepatic, renal, gastrointestinal, ophthalmological, hematologic, neurological, psychiatric, endocrine, immunologic or dermatologic disease
8. Suicidal tendency, history of or disposition to seizures, state of confusion, clinically relevant psychiatric diseases or disorder
9. Presence of out-of-range cardiac interval (PR < 110 msec, PR > 200 msec, QRS < 60 msec, QRS >110 msec and QTc > 440 msec)
10. History of using live attenuated vaccines within 56 days before day 1 of this study
11. Immunization with a vaccine within 28 days before day 1 of this study
12. Use of immunosuppressant in the 28 days before day 1 of this study
13. Maintenance therapy with any drug or significant history of drug dependency or alcohol abuse (> 3 units of alcohol per day, intake of excessive alcohol, acute or chronic)
14. Any clinically significant illness in the previous 28 days before day 1 of this study
15. Use of any enzyme-modifying drugs, including strong inhibitors of cytochrome P450 (CYP) enzymes (such as cimetidine, fluoxetine, quinidine, erythromycin, ciprofloxacin, fluconazole, ketoconazole, diltiazem and HIV antivirals) and strong inducers of CYP enzymes (such as barbiturates, carbamazepine, glucocorticoids, phenytoin, rifampin and St John's Wort), in the previous 28 days before day 1 of this study
16. Any history of latent or active tuberculosis and/or prophylaxis for tuberculosis according to the TB Medical History screening questionnaire (see Appendix 1)
17. Positive tuberculin blood or skin test
18. Herpes IgG (Type 1) and/or IgG (Type 2) antibody levels that may predispose to undesired effects, as per medical judgment
19. Positive urine screening of drugs of abuse
20. Positive alcohol breath test
21. Positive results to HIV Ag/Ab Combo, Hepatitis B surface Antigen (HBsAG (B)(hepatitis B)) or anti-Hepatitis C Virus (HCV (C)) tests
22. Females who are pregnant according to a positive pregnancy test
23. Volunteers who took an Investigational Product (in another clinical trial) with a long half-life (≥120 hours) in the previous 3 months before day 1 of this study
24. Volunteers who took an Investigational Product (in another clinical trial) with a half-life less than 120 hours in the previous 28 days before day 1 of this study or who have already participated in this clinical study
25. Volunteers who donated 50 mL or more of blood in the previous 28 days before day 1 of this study
26. Donation of 500 mL or more of blood (Canadian Blood Services, Hema-Quebec, clinical studies, etc.) in the previous 56 days before day 1 of this study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2015-10-29 (Actual); Primary Completion 2016-01-15 (Actual); Study Completion 2016-01-15 (Actual)

PRIMARY OUTCOMES:
Cmax- Peak Plasma concentration | upto 72 hours
  Peak Plasma concentration of Test product should be comparable with Reference product
AUC0-72 | upto 72 hours
  Area Under the Concentration of Test product should be comparable with Reference product

CONTACTS AND LOCATIONS:
Overall Officials: Eric Sicard, M.D., Principal Investigator — Algorithme Pharma Inc
Locations (1):
- Algorithme Pharma Inc., Mount Royal, Quebec, Canada